CLINICAL TRIAL: NCT04854200
Title: HVAD(TM) SMART 1.0 Study: A Prospective Study of the HVAD(TM) SysteM WAvefoRm and Logfile CharacTeristics
Brief Title: HVAD(TM) SMART 1.0 Study
Status: Withdrawn | Type: Observational
Why Stopped: Product pulled off the market/Production of product stopped
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT19054
Record Dates: First submitted 2021-03-25; First posted 2021-04-22 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Medtronic HeartWare ™ HVAD™ System — The Medtronic HeartWare™ HVAD™ System includes a ventricular assist device (VAD) that helps the heart pump and increases the amount of blood that flows through the body in patients with advanced heart failure.

SUMMARY:
The purpose of HVAD Smart 1.0 study is to collect HVAD device data (i.e., waveform + logfile + pump parameter) in various clinical conditions (e.g., routine follow-up visits, experiencing adverse events) to support development of predictive and actionable algorithms. The collected data will be used to characterize HVAD flow waveform and logfile pattern changes that precede a qualifying adverse event, as well as characterize "normal" HVAD flow waveform and logfile patterns (subjects free from any qualifying adverse event, any hospital readmissions related to a SAE, or any parenteral medical therapy for heart failure management (e.g., inotropes, diuretics, etc.) or ultrafiltration in last 30 days). In addition, the study will collect data to evaluate the utility of CareLink in HVAD patients. The study will not involve any investigational testing and the market-released devices will used as per the approved labelling.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age:
* Refractory, advanced heart failure patient that is either: Prospectively identified as a candidate to receive the commercial HVAD system as their first durable left Ventricular Assist Device (LVAD) implant for approved indications; or within 10 days of receiving the commercial HVAD system as their first durable LVAD for approved indications
* Patient provides written authorization and/or consent per institution and geographical requirements

Exclusion Criteria:

* patient who is, or is expected to be inaccessible for follow up
* patient with previous durable mechanical circulatory support device
* patient with planned Bi-VAD procedure
* patient with exclusion criteria required by local law
* patient is currently enrolled in or plans to enroll in an concurrent drug and/or device study that may confound results (i.e., no required intervention that could affect interpretation of all-around product safety and/or effectiveness). Concomitant observational studies allowed if permitted by IRB/EC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, advanced heart failure patients that meet patient selection criteria for left ventricular assist device (LVAD) implant for any approved indication and implant strategy will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2025-08-22 (Estimated); Study Completion 2025-08-22 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Event Characterization | data collected as events occur throughout study follow-up period; up to the 12 month follow-up visit
  HVAD flow waveform and logfile pattern changes

SECONDARY OUTCOMES:
Qualifying Adverse Event Characterization | data collected as events occur throughout study follow-up period; up to the 12 month follow-up visit
  Measuring HVAD flow waveform and logfile pattern changes for ICVA, HCVA, Pump Thrombosis (PT), GI Bleed, Sepsis, Supraventricular Arrhythmia, Ventricular Arrhythmia, or RHF.
Non-AE/SAE Characterization Group | data collected throughout study follow-up period; up to the 12 month follow-up visit
  Measuring waveform and logfile for subjects in the previous 30 days free from: qualifying AE, hospital readmissions due to SAE, parenteral med therapy for HF management or ultrafiltration.
CareLink Utilization | Up to 12 months post-implant
  Characterizing the utility of CareLink and collect patient outcomes for: rate of unscheduled visits, rate or rehospitalization and length of stay, rate of qualifying AE and HF-related AE's, subject quality of life, and Patient & Physician satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Hayward, M.D., Principal Investigator — Lead PI; Mark S Slaughter, M.D., Principal Investigator — Lead PI

IPD SHARING:
Plan to Share IPD: No